CLINICAL TRIAL: NCT03903484
Title: A Collaborative Intervention for Streamlining Medication Appropriateness and Deprescribing Within Integrated Health-Care Teams
Brief Title: Deprescribing in Primary Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other); Canadian Frailty Network (Other); Horizon Health Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1024257; CAT2017-10 (Other Grant/Funding Number: Canadian Frailty Network)
Record Dates: First submitted 2019-03-27; First posted 2019-04-04 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Inappropriate Prescribing; Primary Health Care; Polypharmacy
Keywords: Frailty; Deprescribing
MeSH Terms: conditions — Frailty | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This is a single group study using a pre-, post-analysis. We will examine medication use, medication appropriateness, quality of life, and satisfaction with the intervention for participants before and after our deprescribing intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deprescribing intervention (Experimental): Included patient participants will meet with their clinical pharmacist to complete a survey about medication use and quality of life. Then working with the pharmacist, patients will prioritize medications that are no longer needed for discontinuing. A deprescribing plan will be created and the pharmacist will work with the patient to complete this plan. The patient will also be provided resources from the study toolbox to support the patients as they work through deprescribing the targeted drugs. Once the deprescribing plan is completed there will be a patient survey that will capture satisfaction with the deprescribing experience and patient quality of life.
  Interventions: Other: Deprescribing toolbox and intervention

INTERVENTIONS:
Other: Deprescribing toolbox and intervention — Pharmacist-led deprescribing plan with the patient which will include the patient's deprescribing goals. The intervention advocates for deprescribing according to recognized algorithms and guidelines which will be included in a resource toolbox/website.

SUMMARY:
Medications can help older adults but can also harm them. Frail older adults tend to have many health problems that require treatment, but are also at risk of harm from the medications prescribed. This makes it hard to get older adults the treatments they need and keep them safe from the harms from medications. It ends up that a lot of visits to emergency rooms and hospitals are due to medications, especially for older adults. Previous research has shown the benefits of stopping medications older adults no longer need. Even so, healthcare professionals do not always do this as well as they could. Our goal is to make a collection of resources for pharmacists who work with doctors and nurses in primary settings that will help support older adults as they safely stop medications that are no longer needed. The investigators will use knowledge and tools that are already known and published. In the first six months the team, which includes older adults and their families, pharmacists, doctors, nurses, and healthcare policymakers developed a framework and resource toolbox that pharmacists can use to help older adults stop medications that are no longer needed. In the remaining 10 months, the investigators will use the resource toolbox in primary healthcare teams and nursing homes. Overall, the investigators expect that by using the resources the pharmacists will be able to support patients stop medications they no longer need and help reduce the number of pills people take, reduce drug costs, reduce harms from medication use and improve quality of life for frail older adults and their loved ones.

DETAILED DESCRIPTION:
As frailty and medical comorbidity increases, the number of medications used increases. The resultant polypharmacy is intended to improve the health status; however, large observational studies refute this premise. In fact, polypharmacy (more than 3 medications) is associated with increased hospitalization (OR 3.79, 95% CI {1.33, 10.90}) and increased mortality (OR 1.27, 95% CI {1.04, 1.56}). With increasing polypharmacy, the risk of adverse health outcomes increases so it is important that deprescribing initiatives are promoted to reduce medication use to improve patient outcomes.

Numerous tools exist that can be used to identify Potentially Inappropriate Medications (PIM), including; Beer's list, STOPP/START, PRISCUS, LAROCHE, Medication Appropriateness Index (MAI), Drug Burden Index, Anticholinergic Drug Scale, Anticholinergic Cognitive Burden Scale, and numerous deprescribing tools from the Canadian Deprescribing Network. The implementation of these tools is not as high as it could or should be, as evidenced by polypharmacy data, such as the 2011 study that found 30% of Canadian seniors aged 65 to 79 took at least five prescription medications concurrently. It is likely that medication use is greater among the oldest old.

The literature is replete with evidence and tools to identify the medications that are the most likely to cause adverse events, however this information is not being translated into practice as medication use and PIM use persists in older adults. Deprescribing is the process of withdrawal of an inappropriate medication supervised by a healthcare professional with the goal of managing polypharmacy and improving outcomes. Healthcare practitioners self-identify that deprescribing is a challenging process. Primary care physicians have increasingly complex patient loads, which contributes to increased numbers of specialist involvement. This makes it challenging to know which medications are necessary and which can be discontinued and whose responsibility it is to initiate and monitor the deprescribing process. In Nova Scotia media has brought attention to PIM use with our high rates of benzodiazepine use. Recent publications have also identified high use of antipsychotics in Nova Scotia.

Previous work suggests including a pharmacist or nurse in deprescribing helps with its success. Indeed, prior work suggests that culture change, and integrated primary care can make a small difference in polypharmacy, but that more targeted interventions with specific engagement of pharmacists is needed. Pharmacists have extensive training in medication use, effects, safety and toxicity. They can identify and resolve medication related issues. Pharmacists can carry out treatment plans in a collaborative environment working with prescribers to monitor medication adherence, effect, and toxicity. Meta-analysis has identified 13 pharmacist led interventions to reduce polypharmacy, which included nine in primary care and two in nursing homes.

Society has a need for improved uptake of deprescribing to support appropriate drug use by adults. The tools and resources available have not led to widespread uptake/implementation. To date deprescribing remains one of the many demands on primary care providers (Family Physicians/Nurse Practitioners). The investigators consider the skill set of pharmacists as ideal to support and monitor patients as they move through the deprescribing process. The investigators recognize that deprescribing cannot happen without extensive communication with primary care providers so that all members of the healthcare team are aware and engaged with the patient and their deprescribing. In considering this collaborative practice clinics with pharmacists embedded in the practice have been identified as sites where pharmacist led deprescribing can successfully support patients through the deprescribing process. This pharmacist led deprescribing process will conform to the standard of care using an evidence supported framework for a selected number of drugs and using recognized deprescribing algorithms and guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Resides in a study long term care facility or visits a study integrated health care clinic;
* Has a general practitioner or nurse practitioner within the team;
* Has stable/good management of any chronic disease that he/she/they has, i.e., the patient has not been hospitalized for the chronic illness within the last three months
* Has not had a change in the targeted medication in the past three months;
* Is taking any drug on the targeted drug list or a drug that the primary care provider and pharmacist agree should be targeted for deprescribing.

Exclusion Criteria:

* Is newly diagnosed (i.e., within the last 6 months) with cancer, stroke, myocardial infarction, diabetes, or chronic obstructive pulmonary disease (COPD), and/or the patient has had a recent surgery (i.e., within the last 6 months);
* Is not able to communicate in English;
* Is end-of-life, as determined by the clinician's professional judgment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Change in patient's medication appropriateness | Before and after deprescribing intervention (counts separated 6 months)
  Change in medication appropriateness index before and after the deprescribing intervention
Healthcare professionals' experience with a collaborative deprescribing intervention | At the end of study (approximately 6 months after the start)
  Mixed methods (qualitative and quantitative) survey measuring satisfaction with deprescribing intervention using a five point Likert scale and open ended questioning.
Change in patient quality of life after deprescribing intervention | Before and after deprescribing intervention (separated 6 months)
  Quality of life survey using EuroQol - 5 Dimension (EQ-5D)
Patient experience with a collaborative deprescribing intervention | Before and after deprescribing intervention (separated 6 months)
  Qualitative post intervention survey

SECONDARY OUTCOMES:
Change in number of medications | Before and after deprescribing intervention (counts separated 6 months)
  The number of medications being used before and after the deprescribing intervention
Change in number of medication administration times per day | Before and after deprescribing intervention (counts separated 6 months)
  The number of times medication are administered in a day before and after the deprescribing intervention
Change in the number of medications used on the anticholinergic cognitive burden scale | Before and after deprescribing intervention (counts separated 6 months)
  The number of medications used on the anticholinergic cognitive burden scale before and after the deprescribing intervention
Change in the number of medications used that are targeted for discontinuation in the intervention | Before and after deprescribing intervention (counts separated 6 months)
  The number of targeted medications used before and after the deprescribing intervention
The number of drugs discontinued | Before and after deprescribing intervention (counts separated 6 months)
  Change in the number of drugs used before and after deprescribing intervention
The number of drugs with doses decreased | Before and after deprescribing intervention (separated 6 months)
  Change in number of drugs with dose decreased that were not discontinued
Decrease in polypharmacy | Before and after deprescribing intervention (counts separated 6 months)
  The number patient participants that were on 5 or more medications before the deprescribing intervention and were on less than 5 medications after the deprescribing intervention
Change in medication cost | Before and after deprescribing intervention (counts separated 6 months)
  Change in medication cost before and after deprescribing intervention
Change in health care utilization | Comparison of the same 6 month period in the preceding year to the 6 month period of the deprescribing intervention
  Number of unplanned hospitalizations
Change in health care utilization | Comparison of the same 6 month period in the preceding year to the 6 month period of the deprescribing intervention
  Number of emergency department visits
Withdrawal reactions as result of deprescribing intervention | During deprescribing intervention (6 months in duration)
  Withdrawal symptoms are discussed at every visit with a healthcare professional and are identified using a general scale (mild, moderate, severe).

CONTACTS AND LOCATIONS:
Overall Officials: Shanna Trennaman, Study Director — Dalhousie University
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia (NS), Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mannucci PM, Nobili A; REPOSI Investigators. Multimorbidity and polypharmacy in the elderly: lessons from REPOSI. Intern Emerg Med. 2014 Oct;9(7):723-34. doi: 10.1007/s11739-014-1124-1. Epub 2014 Aug 28. PMID 25164413
- [Background] Andrew MK, Purcell CA, Marshall EG, Varatharasan N, Clarke B, Bowles SK. Polypharmacy and use of potentially inappropriate medications in long-term care facilities: does coordinated primary care make a difference? Int J Pharm Pract. 2018 Aug;26(4):318-324. doi: 10.1111/ijpp.12397. Epub 2017 Sep 27. PMID 28960614
- [Background] Fried TR, O'Leary J, Towle V, Goldstein MK, Trentalange M, Martin DK. Health outcomes associated with polypharmacy in community-dwelling older adults: a systematic review. J Am Geriatr Soc. 2014 Dec;62(12):2261-72. doi: 10.1111/jgs.13153. PMID 25516023
- [Background] Schottker B, Saum KU, Muhlack DC, Hoppe LK, Holleczek B, Brenner H. Polypharmacy and mortality: new insights from a large cohort of older adults by detection of effect modification by multi-morbidity and comprehensive correction of confounding by indication. Eur J Clin Pharmacol. 2017 Aug;73(8):1041-1048. doi: 10.1007/s00228-017-2266-7. Epub 2017 May 24. PMID 28540438
- [Background] Nossaman VE, Larsen BE, DiGiacomo JC, Manuelyan Z, Afram R, Shukry S, Kang AL, Munnangi S, Angus LDG. Mortality is predicted by Comorbidity Polypharmacy score but not Charlson Comorbidity Index in geriatric trauma patients. Am J Surg. 2018 Jul;216(1):42-45. doi: 10.1016/j.amjsurg.2017.09.011. Epub 2017 Sep 19. PMID 28958648
- [Background] Fastbom J, Johnell K. National indicators for quality of drug therapy in older persons: the Swedish experience from the first 10 years. Drugs Aging. 2015 Mar;32(3):189-99. doi: 10.1007/s40266-015-0242-4. PMID 25673123
- [Background] By the American Geriatrics Society 2015 Beers Criteria Update Expert Panel. American Geriatrics Society 2015 Updated Beers Criteria for Potentially Inappropriate Medication Use in Older Adults. J Am Geriatr Soc. 2015 Nov;63(11):2227-46. doi: 10.1111/jgs.13702. Epub 2015 Oct 8. PMID 26446832
- [Background] O'Mahony D, O'Sullivan D, Byrne S, O'Connor MN, Ryan C, Gallagher P. STOPP/START criteria for potentially inappropriate prescribing in older people: version 2. Age Ageing. 2015 Mar;44(2):213-8. doi: 10.1093/ageing/afu145. Epub 2014 Oct 16. PMID 25324330
- [Background] Holt S, Schmiedl S, Thurmann PA. Potentially inappropriate medications in the elderly: the PRISCUS list. Dtsch Arztebl Int. 2010 Aug;107(31-32):543-51. doi: 10.3238/arztebl.2010.0543. Epub 2010 Aug 9. PMID 20827352
- [Background] Laroche ML, Charmes JP, Merle L. Potentially inappropriate medications in the elderly: a French consensus panel list. Eur J Clin Pharmacol. 2007 Aug;63(8):725-31. doi: 10.1007/s00228-007-0324-2. Epub 2007 Jun 7. PMID 17554532
- [Background] Hanlon JT, Schmader KE, Samsa GP, Weinberger M, Uttech KM, Lewis IK, Cohen HJ, Feussner JR. A method for assessing drug therapy appropriateness. J Clin Epidemiol. 1992 Oct;45(10):1045-51. doi: 10.1016/0895-4356(92)90144-c. PMID 1474400
- [Background] Hilmer SN, Mager DE, Simonsick EM, Cao Y, Ling SM, Windham BG, Harris TB, Hanlon JT, Rubin SM, Shorr RI, Bauer DC, Abernethy DR. A drug burden index to define the functional burden of medications in older people. Arch Intern Med. 2007 Apr 23;167(8):781-7. doi: 10.1001/archinte.167.8.781. PMID 17452540
- [Background] Carnahan RM, Lund BC, Perry PJ, Pollock BG, Culp KR. The Anticholinergic Drug Scale as a measure of drug-related anticholinergic burden: associations with serum anticholinergic activity. J Clin Pharmacol. 2006 Dec;46(12):1481-6. doi: 10.1177/0091270006292126. PMID 17101747
- [Background] Tannenbaum C, Farrell B, Shaw J, Morgan S, Trimble J, Currie J, Turner J, Rochon P, Silvius J. An Ecological Approach to Reducing Potentially Inappropriate Medication Use: Canadian Deprescribing Network. Can J Aging. 2017 Mar;36(1):97-107. doi: 10.1017/S0714980816000702. Epub 2017 Jan 16. PMID 28091333
- [Background] Rotermann M, Sanmartin C, Hennessy D, Arthur M. Prescription medication use by Canadians aged 6 to 79. Health Rep. 2014 Jun;25(6):3-9. PMID 24941315
- [Background] Farrell B, Tsang C, Raman-Wilms L, Irving H, Conklin J, Pottie K. What are priorities for deprescribing for elderly patients? Capturing the voice of practitioners: a modified delphi process. PLoS One. 2015 Apr 7;10(4):e0122246. doi: 10.1371/journal.pone.0122246. eCollection 2015. PMID 25849568
- [Background] Cadogan CA, Ryan C, Francis JJ, Gormley GJ, Passmore P, Kerse N, Hughes CM. Improving appropriate polypharmacy for older people in primary care: selecting components of an evidence-based intervention to target prescribing and dispensing. Implement Sci. 2015 Nov 16;10:161. doi: 10.1186/s13012-015-0349-3. PMID 26573745
- [Background] Anthierens S, Tansens A, Petrovic M, Christiaens T. Qualitative insights into general practitioners views on polypharmacy. BMC Fam Pract. 2010 Sep 15;11:65. doi: 10.1186/1471-2296-11-65. PMID 20840795
- [Background] Trenaman SC, Hill-Taylor BJ, Matheson KJ, Gardner DM, Sketris IS. Antipsychotic Drug Dispensations in Older Adults, Including Continuation After a Fall-Related Hospitalization: Identifying Adherence to Screening Tool of Older Persons' Potentially Inappropriate Prescriptions Criteria Using the Nova Scotia Seniors' Pharmacare Program and Canadian Institute for Health's Discharge Databases. Curr Ther Res Clin Exp. 2018 Aug 31;89:27-36. doi: 10.1016/j.curtheres.2018.08.002. eCollection 2018. PMID 30294400
- [Background] Reeve E, Gnjidic D, Long J, Hilmer S. A systematic review of the emerging de fi nition of 'deprescribing' with network analysis: implications for future research and clinical practice. Br J Clin Pharmacol. 2015 Dec;80(6):1254-68. doi: 10.1111/bcp.12732. PMID 27006985
- [Background] Steinman MA. Polypharmacy-Time to Get Beyond Numbers. JAMA Intern Med. 2016 Apr;176(4):482-3. doi: 10.1001/jamainternmed.2015.8597. No abstract available. PMID 26999383
- [Background] Johansson T, Abuzahra ME, Keller S, Mann E, Faller B, Sommerauer C, Hock J, Loffler C, Kochling A, Schuler J, Flamm M, Sonnichsen A. Impact of strategies to reduce polypharmacy on clinically relevant endpoints: a systematic review and meta-analysis. Br J Clin Pharmacol. 2016 Aug;82(2):532-48. doi: 10.1111/bcp.12959. Epub 2016 May 7. PMID 27059768
- See also: The common pill that's killing in the shadow of the opioid crisis — https://www.cbc.ca/news/canada/nova-scotia/benzodiazepines-opioids-deaths-nova-scotia-1.4937134